CLINICAL TRIAL: NCT06384703
Title: The Evaluation of the Relationship Between Coronary Ectasia And Trimethylamine N Oxide
Brief Title: The Relationship Between Microbiota and Coronary Ectasia
Status: Completed | Type: Observational
Sponsor: Konya Beyhekim Training and Research Hospital (Other Government)
Collaborators: Necmettin Erbakan University (Other)
Responsible Party: Sponsor
Other Study IDs: 201518015
Record Dates: First submitted 2024-04-16; First posted 2024-04-25 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2021-05

CONDITIONS: Coronary Ectasia; Microbial Disease
Keywords: microbiota; endothelium

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — A 3 ml blood sample was taken from the volunteer patients from the femoral artery and radial artery sheath entrance and kept at room temperature for 30 minutes. Then, it was centrifuged at 2500 r.p.m for 15 minutes to obtain a serum sample. The samples obtained within 6 months, which is the collection period of all patients, were stored in Eppendorf tubes at -80 degrees Celsius.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- coronary ectasia cohort: Patients with coronary ectasia detected on coronary angiography and without any exclusion criteria were included.
  Interventions: Diagnostic Test: Taking blood for kit study
- normal coronary cohort: Patients who underwent coronary angiography and did not have any of the exclusion criteria
  Interventions: Diagnostic Test: Taking blood for kit study

INTERVENTIONS:
Diagnostic Test: Taking blood for kit study — Taking blood for kit study (Elisa kit)

SUMMARY:
Introduction: It is now known that the microbiota is far beyond the microbial communities living in certain parts of our body and functions like a metabolic organ. In addition, the microbiota, through its metabolites, is involved in the pathophysiology or progression of a wide range of diseases, from atherosclerotic diseases to metabolic diseases and even neurological diseases. Among these metabolites, trimethylamine n-oxide metabolite has been shown to be particularly effective on atherosclerotic heart diseases.

ELIGIBILITY:
Inclusion Criteria:

* over 18 years old
* not having occlusive coronary artery disease
* having coronary ectasia

Exclusion Criteria:

* patients with chronic kidney disease,
* revascularized coronary artery disease,
* previously documented critical coronary stenosis,
* acute or chronic inflammatory disease,
* rheumatologic disease,
* known active malignant disease,
* heart failure,
* moderate-to-severe valvular pathology
* patients who were on any steroid or immunosuppressive therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: In this study, patients with chronic stable angina who underwent coronary angiography were included after exclusion criteria.
Sampling Method: Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2020-11-03 (Actual); Primary Completion 2021-04-25 (Actual); Study Completion 2021-06-18 (Actual)

PRIMARY OUTCOMES:
death | 1 month
  Death from any cause within the last month

CONTACTS AND LOCATIONS:
Overall Officials: Yakup Alsancak, Principal Investigator — Necmettin Erbakan University
Locations (1):
- Necmettin Erbakan University, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
It was planned to share the trimethylamine N-oxide values obtained from the patients and the basic demographic data of the patients.